CLINICAL TRIAL: NCT01666730
Title: A Phase II Study of Metformin Plus Modified FOLFOX 6 in Patients With Metastatic Pancreatic Cancer
Brief Title: Metformin Plus Modified FOLFOX 6 in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1212
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Metformin; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (metformin hydrochloride, FOLFOX) (Experimental): Patients receive metformin hydrochloride PO BID on days 1-14 and FOLFOX therapy comprising leucovorin calcium IV over 120 minutes, fluorouracil IV continuously over 46 hours, and oxaliplatin IV over 120 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well metformin hydrochloride, leucovorin calcium, fluorouracil, and oxaliplatin work in treating patients with metastatic pancreatic cancer. Metformin hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving metformin hydrochloride together with combination chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if metformin (metformin hydrochloride) when added to FOLFOX ( leucovorin calcium, fluorouracil, oxaliplatin) improves overall survival in patients with metastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. To assess response rate (RR). II. To assess progression free survival (PFS). III. To assess toxicity in patients with metastatic pancreatic cancer receiving FOLFOX and metformin. IV. To identify tumor/serum correlative markers.

OUTLINE: Patients receive metformin hydrochloride orally (PO) twice daily (BID) on days 1-7 for an introductory period before the addition of FOLFOX. After the introductory period, patients will continue metformin twice daily and FOLFOX therapy comprising leucovorin calcium intravenously (IV) over 120 minutes, fluorouracil IV continuously over 46 hours, and oxaliplatin IV over 120 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (or any mixed pathology if adenocarcinoma is predominant)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Patient must have not received systemic chemotherapy for metastatic disease; prior chemotherapy, radiation therapy, concurrent chemoradiation are allowed if used for treatment of non-metastatic disease; prior palliative radiation for symptom management is allowed; any chemotherapy must have been completed 4 weeks prior to enrollment; any radiotherapy must have been completed 2 weeks prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count ≥ 1,500/L
* Platelets ≥ 100,000/L
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Creatinine ≤ 1.5
* Women of childbearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Patients with diabetes are eligible for this trial; all diabetic patients who are enrolled on this study should discuss the need to change their diabetes management regimen with their primary care physician or endocrinologist prior to enrollment
* Diabetic patients who are on metformin are eligible as long as they have been on metformin for less than 6 months (estimated 6 months or less duration of metformin therapy from start of metformin to enrollment on study)

Exclusion Criteria:

* Chemotherapy within 4 weeks prior to entering the study, radiotherapy within 2 weeks prior to entering the study or failure to recover from adverse events due to agents administered more than 4 weeks earlier
* Prior treatment toxicities must be resolved to ≤ grade 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* Current use of metformin for more than 6 months prior to enrollment on study
* Use of any other investigational agents
* Patients with untreated brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biological composition to metformin or oxaliplatin or fluorouracil (5-FU)
* Active second primary malignancy or history of second primary malignancy within the last 3 years, with the exception of basal cell skin cancers or carcinoma in situ that have been adequately treated
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women
* Human immunodeficiency virus (HIV)-positive patients
* Chronic or planned acute alcohol use of three or more drinks per day
* Metabolic acidosis, acute or chronic, including ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bajor, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Started | 50
Completed | 0
Not Completed | 50
Not completed — Adverse Event | 16
Not completed — Death | 2
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 9
Not completed — Disease progression/relapse | 18

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Calculated using Kaplan Meier methods and the median will be estimated assuming an exponential distribution.
Time Frame: Time from first day of treatment to death from any cause, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 50
Months | 7.1 [5.0 to 9.2]

2. Secondary Outcome: Response Rate (RR) Objective Tumor Response Based on Computed Tomography (CT) Scans or Magnetic Resonance Imaging (MRI) Scans According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: CBR is the number of participants of the total analysis population who experience confirmed complete (CR) or partial response (PR) per RECIST
  CR = all detectable tumor has disappeared PR = a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum Stable Disease (SD) = small changes that do not meet previously given criteria. Progressive disease (PD) = a >=20% increase in target lesions
  The true response rate of the combination therapy for this patient population will be estimated based on the number of response using a binomial distribution and its confidence intervals will be estimated using Wilson's method.
Time Frame: 1 year
Population: Patients that were evaluable for clinical response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 31
Participants | 4

3. Secondary Outcome: Clinical Benefit Rate (CBR) Based on Computed Tomography (CT) Scans or Magnetic Resonance Imaging (MRI) Scans According to RECIST
Description: CBR is the number of participants of the total analysis population who experience a CR, PR, or SD per RECIST
  CR = all detectable tumor has disappeared PR = a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum SD = small changes that do not meet previously given criteria. PD = a >=20% increase in target lesions
Time Frame: 1 year
Population: Patients that were evaluable for clinical response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 31
Participants | 14

4. Secondary Outcome: Progression Free Survival According to RECIST 1.1 Criteria
Description: Calculated using Kaplan Meier methods and the median will be estimated assuming an exponential distribution.
Time Frame: Time from first day of treatment received to the earlier documented disease progression or death from any cause, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 50
Months | 5.1 [1.8 to 6.6]

5. Secondary Outcome: Number of Grade 3 and 4 Toxicities According to NCI CTCAE Version 4.0
Description: The toxicity profile of the combination will be tabulated.
Time Frame: Up to 1 year
Measure: Number; unit: Events
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
Number analyzed (Participants) | 50
Events
  Grade 3 | 60
  Grade 4 | 2

ADVERSE EVENTS:
Time Frame: AEs will be collect up to 1 year
Arm/Group | Treatment (Metformin Hydrochloride, FOLFOX)
All-Cause Mortality (participants affected / at risk) | 45/50
Serious Adverse Events (participants affected / at risk) | 9/50
Other Adverse Events (participants affected / at risk) | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Metformin Hydrochloride, FOLFOX) (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1)
Infection- Klebsiella Bacteremia (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Death related to disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Metformin Hydrochloride, FOLFOX) (N=50)
Anemia (Blood and lymphatic system disorders) | 24 (46)
Abdominal pain (Gastrointestinal disorders) | 10 (21)
Bloating (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 13 (18)
Diarrhea (Gastrointestinal disorders) | 17 (32)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 6 (9)
Nausea (Gastrointestinal disorders) | 20 (35)
Vomiting (Gastrointestinal disorders) | 13 (18)
Chills (General disorders) | 4 (4)
Edema limbs (General disorders) | 7 (10)
Fatigue (General disorders) | 28 (59)
Pain (General disorders) | 5 (7)
Mucosal infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (9)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Alanine aminotransferase increased (Investigations) | 10 (12)
Alkaline phosphatase increased (Investigations) | 17 (32)
Aspartate aminotransferase increased (Investigations) | 11 (19)
Blood bilirubin increased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 16 (29)
Neutrophil count decreased (Investigations) | 12 (23)
Platelet count decreased (Investigations) | 17 (38)
Weight loss (Investigations) | 20 (32)
White blood cell decreased (Investigations) | 16 (24)
Dehydration (Metabolism and nutrition disorders) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (30)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (48)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (28)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 13 (26)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (10)
Hyponatremia (Metabolism and nutrition disorders) | 10 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (10)
Dizziness (Nervous system disorders) | 7 (8)
Dysgeusia (Nervous system disorders) | 8 (12)
Paresthesia (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (21)
Anxiety (Psychiatric disorders) | 8 (8)
Depression (Psychiatric disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 14 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT01666730/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT01666730/ICF_001.pdf